CLINICAL TRIAL: NCT03162224
Title: A Phase 1b/2a, Multi-Center Open-Label Study to Evaluate the Safety and Efficacy of Combination Treatment With MEDI0457 (INO-3112) and Durvalumab (MEDI4736) in Patients With Recurrent/Metastatic HPV Associated Head and Neck Squamous Cancer
Brief Title: Safety and Efficacy of MEDI0457 and Durvalumab in Participants With Human Papilloma Virus (HPV) Associated Recurrent/Metastatic Head and Neck Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8860C00005
Record Dates: First submitted 2017-05-15; First posted 2017-05-22 (Actual); Results first posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Head and Neck Cancer; Human Papilloma Virus
Keywords: Head and Neck Squamous Cell Carcinoma; Oropharyngeal Cancer; HPV; Human Papilloma Virus; Cancer Immunotherapy; Check point inhibitors; PD-L1 inhibitor; Recurrent or Metastatic Cancer; Durvalumab; MEDI0457; Antineoplastic agents; Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Oropharyngeal Neoplasms; Recurrence; Neoplasm Metastasis; Neoplasms | interventions — MEDI0457; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- First-line Recurrent/Metastatic (1L R/M) Platinum Non-refractory (Experimental): Participants with recurrent or metastatic disease and were non-refractory to neoadjuvant/adjuvant platinum based chemotherapy, will receive MEDI0457 7 mg intramuscularly followed by electroporation on Day 1 of Weeks 1, 3, 7, 12, and then every 8 weeks (Q8W) and durvalumab 1500 mg intravenously on Day 1 of Week 4 and then every 4 weeks (Q4W) until disease progression, unacceptable toxicity, or withdrawal of consent, whichever occurs first.
  Interventions: Drug: MEDI0457; Device: CELLECTRA®5P device; Drug: Durvalumab
- 1L R/M Platinum Refractory (Experimental): Participants with R/M disease and were refractory to neoadjuvant/adjuvant platinum based chemotherapy, will receive MEDI0457 7 mg intramuscularly followed by electroporation on Day 1 of Weeks 1, 3, 7, 12, and then Q8W and durvalumab 1500 mg intravenously on Day 1 of Week 4 and then Q4W until disease progression, unacceptable toxicity, or withdrawal of consent, whichever occurs first.
  Interventions: Drug: MEDI0457; Device: CELLECTRA®5P device; Drug: Durvalumab
- Second-line (2L) + R/M (Experimental): Participants with R/M disease and were treated with 1 or more lines of platinum based chemotherapy, will receive MEDI0457 7 mg intramuscularly followed by electroporation on Day 1 of Weeks 1, 3, 7, 12, and then Q8W and durvalumab 1500 mg intravenously on Day 1 of Week 4 and then Q4W until disease progression, unacceptable toxicity, or withdrawal of consent, whichever occurs first.
  Interventions: Drug: MEDI0457; Device: CELLECTRA®5P device; Drug: Durvalumab

INTERVENTIONS:
Drug: MEDI0457 — MEDI0457 7 mg will be administered intramuscularly followed by electroporation (EP) using CELLECTRA®5P device.
  Other Names: INO-3112
Device: CELLECTRA®5P device — MEDI0457 7 mg will be administered intramuscularly followed by EP using CELLECTRA®5P device.
  Other Names: CELLECTRA 2000
Drug: Durvalumab — Durvalumab will be administered intravenously at a dose of 1500 mg every 4 weeks.
  Other Names: MEDI4736

SUMMARY:
This is a Phase 1b/2a, open-label, multi-center study to evaluate the safety and tolerability, anti-tumor activity, and immunogenicity of MEDI0457 (also known as INO 3112) a HPV Deoxyribonucleic Acid (DNA) vaccine in combination with durvalumab (also known as MEDI4736) which is a human monoclonal antibody directed against Programmed Death Ligand 1 (PD-L1), which blocks the interaction of PD-L1 with PD-1 and Cluster of differentiation 80 (CD80).

An initial three to 12 participants (Safety Analysis Run-in participants) will be enrolled and assessed for safety before additional participants are enrolled.

The initial safety analysis run-in participants along with an approximate total of 50 participants with human papilloma virus associated recurrent or metastatic head and neck squamous cell cancer (HNSCC) will be enrolled in this study and evaluated also for anti-tumor efficacy to MEDI0457 in combination with durvalumab.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants 18 years and older
2. Histologically or cytologically confirmed diagnosis of HNSCC associated with HPV by a p16 immunohistochemistry (IHC) assay or HPV-16 or HPV-18 positive by nucleic acid testing.
3. Recurrent or metastatic disease that has been treated with at least one platinum-containing regimen and lacking a curative treatment option.
4. Participants who are platinum ineligible may be enrolled if they have received and failed an approved treatment and lack a treatment option with curative potential.

Exclusion criteria:

1. Any concurrent chemotherapy, immune-mediated therapy or biologic or hormonal therapy for cancer treatment Active or prior documented autoimmune disease with some exceptions.
2. Current or prior use of immunosuppressive medication within 14 days prior to first study dose, with the exception of intranasal and inhaled corticosteroids or systemic corticosteroids at doses not to exceed 10 mg/day of prednisone or equivalent. Steroids as premedication for hypersensitivity reactions due to radiographic contrast agents are allowed.
3. No prior exposure to immune-mediated therapy defined as prior exposure to T-cell and natural killer cell directed therapy (e.g., anti-PD-1, anti-PD-L1, anti-CD137, and anti-CTLA4, etc).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MedImmune LLC, Study Director — Study Director
Locations (13):
- United States (13):
  - Research Site, San Francisco, California
  - Research Site, Orlando, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Indianapolis, Indiana
  - Research Site, Baltimore, Maryland
  - Research Site, Detroit, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Morristown, New Jersey
  - Research Site, The Bronx, New York
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: D8860C00005 SAP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8860C00005&attachmentIdentifier=4bf35237-eff1-4bac-9baa-d00fcc13d005&fileName=MEDI_0457_SAP_Main_Body_v4.0_21Jun2021_final_Redacted.pdf&versionIdentifier=
- See also: CSP Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8860C00005&attachmentIdentifier=3b13cfc5-2ea9-489b-bace-19575379de01&fileName=Protocol_Amendment_#8_Actual-Redacted.pdf&versionIdentifier=
- See also: CSR Synopsis Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8860C00005&attachmentIdentifier=d40339f7-44cc-4252-a359-c73c01fe5bf0&fileName=d8860c00005-abbreviated-study-synopsis_100322-Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The data are reported per the data cut-off (DCO) date of 19Mar2021 and the data after DCO will not be entered into the clinical study database and hence, will not be analyzed.
Groups:
- First-line Recurrent/Metastatic (1L R/M) Platinum Non-refractory: Participants with recurrent or metastatic disease and were non-refractory to neoadjuvant/adjuvant platinum based chemotherapy, received MEDI0457 7 mg intramuscularly followed by electroporation on Day 1 of Weeks 1, 3, 7, 12, and then every 8 weeks (Q8W) and durvalumab 1500 mg intravenously on Day 1 of Week 4 and then every 4 weeks (Q4W) until disease progression, unacceptable toxicity, or withdrawal of consent, whichever occurred first.
- 1L R/M Platinum Refractory: Participants with R/M disease and were refractory to neoadjuvant/adjuvant platinum based chemotherapy, received MEDI0457 7 mg intramuscularly followed by electroporation on Day 1 of Weeks 1, 3, 7, 12, and then Q8W and durvalumab 1500 mg intravenously on Day 1 of Week 4 and then Q4W until disease progression, unacceptable toxicity, or withdrawal of consent, whichever occurred first.
- Second-line (2L) + R/M: Participants with R/M disease and were treated with 1 or more lines of platinum based chemotherapy, received MEDI0457 7 mg intramuscularly followed by electroporation on Day 1 of Weeks 1, 3, 7, 12, and then Q8W and durvalumab 1500 mg intravenously on Day 1 of Week 4 and then Q4W until disease progression, unacceptable toxicity, or withdrawal of consent, whichever occurred first.
Period: Overall Study
Arm/Group | First-line Recurrent/Metastatic (1L R/M) Platinum Non-refractory | 1L R/M Platinum Refractory | Second-line (2L) + R/M
Started | 15 | 9 | 11
Completed | 4 | 1 | 1
Not Completed | 11 | 8 | 10
Not completed — Death | 4 | 5 | 8
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Other | 6 | 2 | 1

BASELINE CHARACTERISTICS:
Population: As-treated population included all participants who received at least one dose of any study drug.
Groups:
- 1L R/M Platinum Non-refractory: Participants with recurrent or metastatic disease and were non-refractory to neoadjuvant/adjuvant platinum based chemotherapy, received MEDI0457 7 mg intramuscularly followed by electroporation on Day 1 of Weeks 1, 3, 7, 12, and then Q8W and durvalumab 1500 mg intravenously on Day 1 of Week 4 and then Q4W until disease progression, unacceptable toxicity, or withdrawal of consent, whichever occurred first.
- 2L+R/M: Participants with R/M disease and were treated with 1 or more lines of platinum based chemotherapy, received MEDI0457 7 mg intramuscularly followed by electroporation on Day 1 of Weeks 1, 3, 7, 12, and then Q8W and durvalumab 1500 mg intravenously on Day 1 of Week 4 and then Q4W until disease progression, unacceptable toxicity, or withdrawal of consent, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | 1L R/M Platinum Non-refractory | 1L R/M Platinum Refractory | 2L+R/M | Total
Number analyzed (Participants) | 15 | 9 | 11 | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.6 (8.60) | 57.3 (7.98) | 60.4 (5.28) | 61.0 (7.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 1
  Male | 15 | 8 | 11 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 9 | 11 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 0 | 1 | 0 | 1
  White | 15 | 7 | 11 | 33
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug. There will be no updated results for this outcome measures at the time of end of study.
Time Frame: Day 1 through 90 days after the last dose of study drug (approximately 45 months)
Population: As-treated population included all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 1L R/M Platinum Non-refractory | 1L R/M Platinum Refractory | 2L+R/M
Number analyzed (Participants) | 15 | 9 | 11
Participants
  Any TEAE | 15 | 9 | 11
  Any TESAE | 4 | 4 | 6

2. Primary Outcome: Number of Participants With Abnormal Laboratory Parameters Reported as TEAEs
Description: Any laboratory abnormality during analysis of hematology, clinical chemistry, thyroid function tests, and urinalysis that was new in onset or worsened in severity or frequency from the baseline condition and required therapeutic intervention or diagnostic tests, led to discontinuation of study treatment, had accompanying or inducing symptoms or signs, or judged by the Investigator as clinically significant was recorded as AE. Participants with abnormal laboratory parameters reported as TEAEs are reported.
Time Frame: Day 1 through 90 days after the last dose of study drug (approximately 45 months)
Population: As-treated population included all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 1L R/M Platinum Non-refractory | 1L R/M Platinum Refractory | 2L+R/M
Number analyzed (Participants) | 15 | 9 | 11
Participants
  Lymphocyte count decreased | 2 | 1 | 3
  Aspartate aminotransferase increased | 1 | 1 | 3
  Alanine aminotransferase increased | 2 | 1 | 1
  Lipase increased | 2 | 1 | 1
  Neutrophil count decreased | 1 | 1 | 1
  Platelet count decreased | 2 | 1 | 0
  White blood cell count decreased | 1 | 1 | 1
  Blood creatinine increased | 1 | 1 | 0
  Blood thyroid stimulating hormone increased | 0 | 1 | 1
  Blood urea increased | 2 | 0 | 0
  Amylase increased | 0 | 0 | 1
  Blood alkaline phosphatase increased | 0 | 0 | 1
  Blood bilirubin increased | 0 | 1 | 0
  Blood creatine phosphokinase increased | 0 | 0 | 1
  Red blood cell count decreased | 1 | 0 | 0
  Tri-iodothyronine decreased | 0 | 1 | 0
  Troponin T increased | 1 | 0 | 0
  White blood cell count increased | 0 | 1 | 0
  Hyponatraemia | 1 | 3 | 2
  Hyperglycaemia | 3 | 1 | 1
  Hypokalaemia | 0 | 3 | 1
  Hypoalbuminaemia | 0 | 0 | 2
  Hypomagnesaemia | 0 | 1 | 1
  Hypocalcaemia | 0 | 0 | 1
  Hypoglycaemia | 0 | 1 | 0
  Hypophosphataemia | 0 | 1 | 0
  Hypothyroidism | 3 | 2 | 2
  Hyperthyroidism | 0 | 1 | 2
  Anaemia | 3 | 5 | 4
  Neutropenia | 0 | 1 | 0
  Lymphopenia | 0 | 0 | 1

3. Primary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Reported as TEAEs
Description: Participants with ECG abnormalities reported as TEAEs are reported.
Time Frame: Day 1 through 90 days after the last dose of study drug (approximately 45 months)
Population: As-treated population included all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 1L R/M Platinum Non-refractory | 1L R/M Platinum Refractory | 2L+R/M
Number analyzed (Participants) | 15 | 9 | 11
Participants
  Atrial fibrillation | 1 | 2 | 1
  Bradycardia | 0 | 0 | 3
  Sinus tachycardia | 1 | 1 | 1
  Sinus bradycardia | 1 | 1 | 0
  Cardiac failure | 1 | 0 | 0
  Left ventricular hypertrophy | 0 | 1 | 0
  Myocarditis | 1 | 0 | 0
  Pericardial effusion | 0 | 1 | 0
  Supraventricular tachycardia | 0 | 1 | 0

4. Primary Outcome: Number of Participants With Abnormal Vital Signs and/or Physical Examination Reported as TEAEs
Description: Vital sign assessment included body temperature, respiration rate, pulse oximetry, blood pressure, heart rate, and weight. Participants with abnormal vital sign and/or abnormal physical examination reported as TEAEs are reported.
Time Frame: Day 1 through 90 days after the last dose of study drug (approximately 45 months)
Population: As-treated population included all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 1L R/M Platinum Non-refractory | 1L R/M Platinum Refractory | 2L+R/M
Number analyzed (Participants) | 15 | 9 | 11
Participants
  Pyrexia | 1 | 4 | 2
  Weight decreased | 4 | 2 | 2
  Weight increased | 2 | 0 | 0
  Breath sounds abnormal | 0 | 0 | 1
  Dyspnoea | 4 | 4 | 3
  Hypertension | 5 | 1 | 4
  Hypotension | 1 | 0 | 2
  Blood pressure increased | 1 | 0 | 0

5. Primary Outcome: Number of Participants Who Received Any Concomitant Medications During the Study
Description: Participants who received concomitant medications which were ongoing at the start of treatment or started after the study treatment are included.
Time Frame: Day 1 through 90 days after the last dose of study drug (approximately 45 months)
Population: As-treated population included all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 1L R/M Platinum Non-refractory | 1L R/M Platinum Refractory | 2L+R/M
Number analyzed (Participants) | 15 | 9 | 11
Participants | 15 | 9 | 11

6. Primary Outcome: Number of Participants With Shift >=3 Changed From Baseline in Eastern Cooperative Oncology Group Performance (ECOG) Status
Description: Participants with shift >=3 changed from baseline in ECOG status are reported. ECOG performance status is used by doctors and researchers to assess how a participant's disease is progressing, assess how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis. The scores are: 0 = Fully Active, able to carry out all pre-disease performance without restrictions; 1 = Restricted activity but ambulatory and able to carry out light work or work of a sedentary nature; 2 = Ambulatory and capable of self-care but unable to carry out work activities; 3 = Capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4 = Completely Disabled, unable to carry out any self-care and totally confined to bed or chair; 5 = Dead.
Time Frame: Day 1 through 90 days after the last dose of study drug (approximately 45 months)
Population: As-treated population included all participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 1L R/M Platinum Non-refractory | 1L R/M Platinum Refractory | 2L+R/M
Number analyzed (Participants) | 15 | 9 | 11
Participants | 0 | 0 | 1

7. Primary Outcome: Percentage of Participants With Objective Response by Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 in Response-evaluable Population
Description: The objective response is defined as confirmed complete response (CR) or confirmed partial response (PR) based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) guidelines. The CR is defined as disappearance of all target and non-target lesions, no new lesions, and normalization of tumor marker level. The PR is defined as >= 30% decrease in the sum of the diameters of target lesions compared to baseline and no new non-target lesion. A confirmed CR or PR is defined as 2 CRs or 2 PRs that were separated by at least 4 weeks with no evidence of progression or not evaluable response in-between. Percentage of participants with objective response is reported.
Time Frame: Day 1 through end of study (approximately 45 months)
Population: Response-evaluable population included all participants with confirmed human papilloma virus Type 16 (HPV-16) or HPV-18 associated disease, who received one dose of both study drugs, had a baseline scan (Days -28 to -1) with measurable disease at baseline, and at least one follow-up scan with the opportunity to be followed for >= 16 weeks.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 1L R/M Platinum Non-refractory | 1L R/M Platinum Refractory | 2L+R/M
Number analyzed (Participants) | 12 | 7 | 10
Percentage of participants | 33.3 [9.92 to 65.11] | 28.6 [3.67 to 70.96] | 20.0 [5.73 to 43.66]

8. Secondary Outcome: Percentage of Participants With Objective Response by RECIST Version 1.1 in As-treated Population
Description: The objective response is defined as confirmed CR or confirmed PR based on RECIST v1.1 guidelines. The CR is defined as disappearance of all target and non-target lesions, no new lesions, and normalization of tumor marker level. The PR is defined as >= 30% decrease in the sum of the diameters of target lesions compared to baseline and no new non-target lesion. A confirmed CR or PR is defined as 2 CRs or 2 PRs that were separated by at least 4 weeks with no evidence of progression or not evaluable response in-between. Percentage of participants with objective response is reported.
Time Frame: Day 1 through end of study (approximately 45 months)
Population: As-treated population included all participants who received at least one dose of any study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 1L R/M Platinum Non-refractory | 1L R/M Platinum Refractory | 2L+R/M
Number analyzed (Participants) | 15 | 9 | 11
Percentage of participants | 33.3 [11.82 to 61.62] | 22.2 [2.81 to 60.01] | 18.2 [5.19 to 40.28]

9. Secondary Outcome: Percentage of Participants With Objective Response by Immune-related RECIST (irRECIST) in Response-evaluable Population
Description: The objective response is defined as confirmed CR or confirmed PR based on irRECIST v1.1 guidelines. The irCR is defined as disappearance of all target and non-target lesions, no new lesions, and normalization of tumor marker level. The irPR is defined as >= 50% decrease in the sum of the diameters of target lesions compared to baseline and no new non-target lesion. A confirmed irCR or irPR is defined as 2 irCRs or 2 irPRs that were separated by at least 4 weeks with no evidence of progression or not evaluable response in-between. Percentage of participants with objective response is reported.
Time Frame: Day 1 through end of study (approximately 45 months)
Population: Response-evaluable population included all participants with confirmed HPV-16 or HPV-18 associated disease, who received one dose of both study drugs, had a baseline scan (Days -28 to -1) with measurable disease at baseline, and at least one follow-up scan with the opportunity to be followed for >= 16 weeks.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 1L R/M Platinum Non-refractory | 1L R/M Platinum Refractory | 2L+R/M
Number analyzed (Participants) | 12 | 7 | 10
Percentage of participants | 41.7 [15.17 to 72.33] | 28.6 [3.67 to 70.96] | 20.0 [2.52 to 55.61]

10. Secondary Outcome: Percentage of Participants With Objective Response by irRECIST in As-treated Population
Description: as for outcome 9
Time Frame: Day 1 through end of study (approximately 45 months)
Population: As-treated population included all participants who received at least one dose of any study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 1L R/M Platinum Non-refractory | 1L R/M Platinum Refractory | 2L+R/M
Number analyzed (Participants) | 15 | 9 | 11
Percentage of participants | 40.0 [16.34 to 67.71] | 22.2 [2.81 to 60.01] | 18.2 [2.28 to 51.78]

11. Secondary Outcome: Disease Control Rate (DCR) at Week 16 by RECIST Version 1.1 in Response-evaluable Population
Description: The DCR is defined percentage of participants with CR, PR, or stable disease (SD) at 16 weeks based on RECIST v1.1 guidelines. A CR is defined as disappearance of all target and non-target lesions, no new lesions, and normalization of tumor marker level. A PR is defined as >= 30% decrease in the sum of longest diameters of target lesions compared to baseline and no new non-target lesion. The SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression, taking as reference the smallest sum longest diameter since the study treatment started, and persistence of one or more non-target lesion(s) or / and maintenance of tumor marker level above the normal limits.
Time Frame: Week 16
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 1L R/M Platinum Non-refractory | 1L R/M Platinum Refractory | 2L+R/M
Number analyzed (Participants) | 12 | 7 | 10
Percentage of participants | 50.0 [21.09 to 78.91] | 28.6 [3.67 to 70.96] | 50.0 [27.20 to 72.80]

12. Secondary Outcome: DCR at Week 16 by RECIST Version 1.1 in As-treated Population
Description: The DCR is defined percentage of participants with CR, PR, or SD at 16 weeks based on RECIST v1.1 guidelines. A CR is defined as disappearance of all target and non-target lesions, no new lesions, and normalization of tumor marker level. A PR is defined as >= 30% decrease in the sum of longest diameters of target lesions compared to baseline and no new non-target lesion. The SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression, taking as reference the smallest sum longest diameter since the study treatment started, and persistence of one or more non-target lesion(s) or / and maintenance of tumor marker level above the normal limits.
Time Frame: Week 16
Population: As-treated population included all participants who received at least one dose of any study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 1L R/M Platinum Non-refractory | 1L R/M Platinum Refractory | 2L+R/M
Number analyzed (Participants) | 15 | 9 | 11
Percentage of participants | 53.3 [26.59 to 78.73] | 33.3 [7.49 to 70.07] | 45.5 [24.39 to 67.79]

13. Secondary Outcome: Progression Free Survival (PFS)
Description: The PFS is defined as the time from the date of start of study treatment until the documentation of disease progression based on RECIST version 1.1 or death due to any cause, whichever occurs first. The progressive disease is defined at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started, the appearance of one or more new lesions, or unequivocal progression of existing non-target lesions. Participants who were not progressed or died at the time of the analysis were censored at the time of the latest date of assessment from their last evaluable RECIST version 1.1 assessment. The PFS was estimated using Kaplan-Meier method.
Time Frame: Day 1 through end of study (approximately 45 months)
Population: As-treated population included all participants who received at least one dose of any study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 1L R/M Platinum Non-refractory | 1L R/M Platinum Refractory | 2L+R/M
Number analyzed (Participants) | 15 | 9 | 11
Months | 9.5 [1.88 to NA] — Upper limit of 95% Confidence Interval (CI) was not reached because an insufficient number of participants had PFS. | 2.3 [0.63 to NA] — Upper limit of 95% CI was not reached because an insufficient number of participants had PFS. | 3.8 [1.68 to 5.63]

14. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from the date of start of study treatment until death due to any cause. Any participant not died at the time of analysis was censored based on the last recorded date on which the participant was known to be alive. The OS was estimated using Kaplan-Meier method.
Time Frame: Day 1 through end of study (approximately 45 months)
Population: As-treated population included all participants who received at least one dose of any study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 1L R/M Platinum Non-refractory | 1L R/M Platinum Refractory | 2L+R/M
Number analyzed (Participants) | 15 | 9 | 11
Months | NA [13.62 to NA] — Median and upper limit of 95% CI were not reached because an insufficient number of participants had OS. | 29.2 [0.63 to NA] — Upper limit of 95% CI was not reached because an insufficient number of participants had OS. | 19.2 [14.84 to 26.97]

15. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibodies (ADA) to Durvalumab
Description: Number of participants with positive ADA titer to durvalumab are reported. ADA prevalence is defined as ADA positive at any point (baseline and post-baseline); persistent positive is defined as ADA positive at Week 16, and transient positive is defined as positive at Week 8 but not at Week 16, regardless of baseline positivity.
Time Frame: Pre-dose (up to 60 minutes prior to durvalumab administration) on Week 4, Week 8, and Week 16
Population: The ADA evaluable population included all participants who had non-missing baseline ADAs (on Day 1) and at least one non-missing post-baseline ADA result.
Measure: Count of Participants; unit: Participants
Arm/Group | 1L R/M Platinum Non-refractory | 1L R/M Platinum Refractory | 2L+R/M
Number analyzed (Participants) | 15 | 9 | 11
Participants
  ADA prevalence | 0 | 0 | 1
  Persistent positive ADA | 0 | 0 | 0
  Transient positive ADA | 0 | 0 | 0

16. Secondary Outcome: Serum Concentrations of Durvalumab
Description: Serum concentrations of durvalumab is reported.
Time Frame: Pre-dose (up to 60 minutes prior to durvalumab administration) on Week 4, Week 8, and Week 16
Population: Pharmacokinetics population included all participants who received at least one dose of durvalumab and had at least one evaluable post-dose serum concentration measurement of durvalumab. 'Number analyzed' denotes the number of participants evaluated for the specified time point.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | 1L R/M Platinum Non-refractory | 1L R/M Platinum Refractory | 2L+R/M
Number analyzed (Participants) | 12 | 7 | 10
mg/L
  Week 4 pre-dose: number analyzed (Participants) | 1 | 1 | 0
  Week 4 pre-dose | 0.767 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified time point. | 1.505 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified time point. |
  Week 8 pre-dose | 92.163 (37.823) | 89.094 (69.586) | 94.665 (50.546)
  Week 16 pre-dose: number analyzed (Participants) | 10 | 4 | 5
  Week 16 pre-dose | 190.061 (94.466) | 127.269 (56.927) | 121.728 (79.189)

ADVERSE EVENTS:
Time Frame: Day 1 through 90 days after the last dose of study drug (approximately 45 months)
Groups:
- 1L R/M Platinum Non-refractory; 1L R/M Platinum Refractory; 2L+ R/M: Description (Arm-group)
Arm/Group | 1L R/M Platinum Non-refractory | 1L R/M Platinum Refractory | 2L+ R/M
All-Cause Mortality (participants affected / at risk) | 4/15 | 5/9 | 8/11
Serious Adverse Events (participants affected / at risk) | 4/15 | 4/9 | 6/11
Other Adverse Events (participants affected / at risk) | 15/15 | 9/9 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1L R/M Platinum Non-refractory (N=15) | 1L R/M Platinum Refractory (N=9) | 2L+ R/M (N=11)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1L R/M Platinum Non-refractory (N=15) | 1L R/M Platinum Refractory (N=9) | 2L+ R/M (N=11)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Incision site erythema (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Nasal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Osteoradionecrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (3) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Deafness bilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 5 (7) | 4 (8)
Hypothyroidism (Endocrine disorders) | 3 (3) | 2 (2) | 2 (2)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Corneal thinning (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 1 (2)
Retinal tear (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (5) | 2 (6) | 2 (9)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Lip dry (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5) | 2 (4) | 3 (3)
Salivary hypersecretion (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (4) | 1 (1)
Administration site bruise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Administration site induration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Administration site pain (General disorders) | 2 (7) | 1 (2) | 1 (8)
Administration site reaction (General disorders) | 1 (1) | 1 (1) | 0 (0)
Administration site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Catheter site pruritus (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (3)
Chills (General disorders) | 2 (2) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 1 (2) | 1 (1)
Facial pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 9 (16) | 6 (6) | 4 (4)
Fibrosis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site discomfort (General disorders) | 1 (2) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 4 (12) | 4 (13) | 1 (1)
Injection site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (3) | 1 (1) | 1 (2)
Non-cardiac chest pain (General disorders) | 3 (4) | 0 (0) | 2 (3)
Oedema peripheral (General disorders) | 2 (2) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 4 (4) | 2 (2)
Swelling face (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vaccination site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Epididymitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 1 (3) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Oral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pilonidal cyst (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (2) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (5) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (3) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (3)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 1 (1) | 1 (2)
Blood urea increased (Investigations) | 2 (3) | 0 (0) | 0 (0)
Breath sounds abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 2 (2) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (7) | 1 (3) | 3 (7)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Platelet count decreased (Investigations) | 2 (3) | 1 (1) | 0 (0)
Red blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Tri-iodothyronine decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Troponin t increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 4 (4) | 2 (3) | 2 (6)
Weight increased (Investigations) | 2 (3) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1) | 1 (2)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 1 (6)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (6) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 3 (5) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (11) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (4) | 4 (4)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (5) | 1 (2) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (6) | 3 (5)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 1 (1)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Accessory nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (3) | 2 (2)
Dizziness postural (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 3 (4) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle spasticity (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vertebral artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Device leakage (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (4) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0) | 2 (2)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Scrotal erythema (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 4 (6) | 7 (8)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (5) | 3 (4)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 1 (1) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 1 (1)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (4) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (8) | 2 (4) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Reactive perforating collagenosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 5 (8) | 1 (3) | 4 (11)
Hypotension (Vascular disorders) | 1 (2) | 0 (0) | 2 (2)
Lymphoedema (Vascular disorders) | 1 (1) | 1 (1) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 2 (3) | 2 (2)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mouth swelling (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The expected response in terms of efficacy was not achieved at the time of DCO. It was therefore decided to stop further enrollment of participants and the study was terminated. There were no safety concerns were noted with the combination of MEDI0457 and durvalumab.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/24/NCT03162224/Prot_002.pdf
  • Statistical Analysis Plan (2021-06-21): https://cdn.clinicaltrials.gov/large-docs/24/NCT03162224/SAP_003.pdf